CLINICAL TRIAL: NCT03720600
Title: Examination of a Mindfulness- and Acceptance-Based Health Promotion Program on Momentary Experiences of Racism and Mental Health Outcomes
Brief Title: Forms of Racial Discrimination Study
Acronym: FORD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jennifer Martinez, Doctoral Candidate, University of Massachusetts, Boston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018026; 1R36MH116678-01 (NIH)
Record Dates: First submitted 2018-10-22; First posted 2018-10-25 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Psychological Distress
Keywords: mindfulness; acceptance; racism
MeSH Terms: conditions — Racism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MAB Intervention (Experimental): Participants in this condition will be asked to come into the laboratory twice. At Time 1 (T1), participants in this condition will watch a voice-guided PowerPoint on MAB strategies for coping with discrimination. For the following two weeks, they will be asked to complete multiple momentary assessments daily for two weeks. After two weeks, participants will return to the laboratory to complete a final battery of questionnaires and complete a qualitative exit-interview.
  Interventions: Behavioral: MAB Intervention
- Waitlist-Control (Other): Participants in the "waitlist-control" condition will be asked to come into the laboratory twice. At Time 1 (T1), participants in this condition will complete an initial set of questionnaires. For the following two weeks, they will be asked to complete multiple daily momentary assessments daily. After two weeks, participants will return to the laboratory to complete a final battery of questionnaires, watch a voice-guided PowerPoint on MAB strategies for coping with discrimination, and complete a qualitative exit-interview.
  Interventions: Behavioral: MAB Intervention
- No-EMA Control (No Intervention): Participants in the "No-EMA Control" condition will only complete questionnaires at T1 and T2.

INTERVENTIONS:
Behavioral: MAB Intervention — The intervention is a 60-minute voice-recorded PowerPoint presentation on a mindfulness- and acceptance-based (MAB) intervention adapted from Eustis et al. (2017). This adaptation was informed by research on MAB therapies and other approaches to coping with discrimination (e.g., Watson, Black, & Hunter, 2016), as well as clinical experience providing an in-person workshop on MAB strategies for coping with racism-related stress.
  Arms: MAB Intervention; Waitlist-Control

SUMMARY:
The project aims to evaluate a brief intervention for coping with racism-related experiences for people of color and examine momentary factors that may buffer the negative mental health impact of racism.

DETAILED DESCRIPTION:
This study focuses on the unique experiences of people of color (e.g., Asian American, Black/African American, Latinx, Native, Multiracial), ways they manage coping with race-related stress, as well as evaluating the effectiveness of a brief, one-hour intervention focused on coping with racism. First, the study will evaluate the acceptability and impact of a brief, single-session, 1-hour intervention aimed at addressing strategies for coping with racism compared to a waitlist-control condition. The intervention will integrate culturally-adapted approaches for enhancing compassionate awareness, emotional acceptance, valued actions, and coping flexibility (CAAVAF). The study will also evaluate whether the brief CAAVAF program will be associated with increased use of CAAVAF strategies (compassionate awareness, emotional acceptance, valued action, and coping flexibility) in response to racial discrimination over time and whether the brief CAAVAF program improves mental health outcomes at the two-week follow-up. Second, the study aims to evaluate the impact of CAAVAF strategies on mental health outcomes in response to momentary reports of coping with discrimination and from pre- to two-week follow-up.

All participants will be asked to complete an online screening questionnaire, which will include informed consent, demographic questionnaires, past experiences of discrimination, and trait measures of coping. Participants will be randomized into a.) a CAAVAF program, b.) a waitlist control condition with EMA, or c.) a control condition without the CAAVAF program or EMA. Participants in the CAAVAF condition will watch a scripted CAAVAF psychoeducation video during an initial laboratory session; in contrast, participants in the waitlist control condition will watch the video in a second session (after two weeks of ecological momentary assessment). Participants in both the CAAVAF program and waitlist control condition will be given instructions on using an EMA cellphone application during the initial session for repeated momentary assessments. Following this session, participants in the EMA conditions will monitor their experiences of discrimination over two weeks, and report their mood and strategies used. Participants will then return to the lab and complete a final battery of questionnaires and a qualitative exit-interview. Participants in the control condition will only complete pre questionnaires and questionnaires at a two-week follow-up.Study findings will contribute to the existing literature by evaluating whether CAAVAF strategies are effective buffers against racism-related mental health outcomes, and whether our CAAVAF and EMA program facilitates the use of these strategies.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as a person of color (not white, European American)
* self-reported distress from racial microaggressions (score of 24 or higher on the Racial Microaggressions Scale; this score is 1 SD deviation below the mean in an unpublished dataset from a study conducted at the same institution)

Exclusion Criteria:

* Has lived in the U.S. for less than 5 years
* Not fluent in English
* Identifies as White, European American

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Depression Anxiety and Stress Scale scores | Baseline and two weeks later
  21-item self-report measure of past-week depressive and anxious symptoms. Each item is rated on a 4-point Likert scale (0= Did not apply to me at all, to 3= Applied to me very much or most of the time). Subscale scores are summed, with higher scores indicating more persistent depressive or anxious symptoms.

SECONDARY OUTCOMES:
Momentary changes in Positive And Negative Affect Scale | four times a day for two weeks
  20-item self-report measure of positive and negative emotions at the present moment. Each item is rated on a 5-point Likert scale (1=very slightly or not at all to 5=extremely). Subscale scores are summed, with higher scores indicating greater positive or negative affect.
Quantitative measure of intervention helpfulness | Two weeks after baseline
  8-item measure developed by PI and colleagues to assess intervention helpfulness. Items are rated on a 5-point Likert scale (1=extremely unhelpful/not at all helpful to 5=extremely helpful/definitely helpful). Items will be summed, with higher scores indicating greater reports of helpfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer H. Martinez, M.A., Principal Investigator — University of Massachusetts, Boston
Locations (1):
- University of Massachusetts Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will include data from approximately 100 subjects who will complete a coping with racism health promotion program and two-week momentary assessments at an urban university. The final dataset will include self-reported demographic, mood, and behavioral data from online questionnaires.
Supporting Information: Study Protocol, ICF, CSR